CLINICAL TRIAL: NCT06837376
Title: Effects of Metabolic Testing Data and Education on Attitudes and Beliefs Related to Carbohydrate Intake in Adolescent Female Athletes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-2408
Record Dates: First submitted 2025-02-14; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Nutritional Deficiency
Keywords: exercise performance; metabolic testing; education; carbohydrate; adolescent; female; athlete
MeSH Terms: conditions — Malnutrition | interventions — Educational Status; Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education plus metabolic testing (Other): Classroom session with slides and videos. Exercise with shared exercise data.
  Interventions: Other: Education; Other: Metabolic Testing (Exercise) with shared interpreted results
- Education only (Other): Classroom session with slides and videos.
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — One 45 minute educational session on the role of carbohydrate in exercise
Other: Metabolic Testing (Exercise) with shared interpreted results — One 20-30 minute session. Treadmill, warm-up, then at increasing intensities for 3-minute intervals wearing a mouthpiece for measurement of respiratory gasses (oxygen consumption, carbon dioxide production). Testing starts with a 3-minute warm-up at 3.4 mph, 1% grade, increasing every 3 minutes until a respiratory exchange ratio of 1.0 is reached or volitional exhaustion
  Arms: Education plus metabolic testing

SUMMARY:
Many studies have consistently shown that females across sports under consume carbohydrate. Registered dietitians working with athletes have also reported female athletes chronically under consume carbohydrate. The primary objective of this study is to compare the effectiveness of education versus education plus interpreted individual metabolic (exercise) testing results to change attitudes and beliefs of female athletes regarding carbohydrate intake. The secondary objective is to assess the effectiveness of the education alone on attitudes and beliefs towards consuming carbohydrate in female athletes.

The study hypothesis is that education alone will not significantly impact attitudes and beliefs, and that metabolic testing and the interpretation of the individual results will alter attitudes and beliefs toward carbohydrate intake.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged between the ages of 13-19 years old
2. Non-smoker
3. Currently enrolled in an IMG Academy sport
4. Willing to fast overnight (10 hours) prior to testing (for metabolic testing group).
5. Understand the protocol and be able to give verbal and written informed consent for participation as well as obtain parental consent if <18 years of age.
6. Must be fluent in English reading, writing, and speaking.
7. You are not employed by, or have a parent, guardian, or other immediate family member employed by a company that manufactures any products that compete with any Gatorade product. If you are unsure if a company would be considered a competitor to Gatorade, let the study investigator know the name of the other company and the nature of your relationship to that company before you sign the informed consent
8. If subject has asthma, they may still participate in but will be required to bring their prescribed inhaler if placed in the metabolic testing group

Exclusion Criteria:

1. Expulsion from school for any reason
2. Leaving the IMG sports team
3. Pregnant or planning to become pregnant
4. Participated in any other clinical trial in the past 30 day
5. Participated in any PepsiCo trial in the past 6 months
6. Physical injury that would prevent participation in exercise group

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Education versus Education plus metabolic testing | Change in Nutrition Attitudes Questionnaire score from Baseline visit to same questionnaire re-taken 2 weeks later. For each questionnaire, a higher score will be correlated to more positive sentiments around carbohydrate intake.
  To compare the effectiveness of education alone versus education plus interpreted individual metabolic testing results to change attitudes and beliefs of female athletes regarding carbohydrate intake.

SECONDARY OUTCOMES:
Education alone | Change in Nutrition Attitudes Questionnaire score from Baseline visit to same questionnaire re-taken 2 weeks later. A higher score will be correlated to more positive sentiments around carbohydrate intake.
  Within the education only group

CONTACTS AND LOCATIONS:
Overall Officials: Kris Osterberg, PhD, RD, Principal Investigator — PepsiCo R&D Life Sciences, Sports Science
Locations (1):
- Gatorade Sports Science Institute at IMG Academy, Bradenton, Florida, United States

IPD SHARING:
Plan to Share IPD: No